CLINICAL TRIAL: NCT01138189
Title: A Prospective Eye to Eye Comparison of LASIK Using Wavefront-guided Treatment Versus Wavefront-optimized Treatment
Brief Title: Wavefront-guided Versus Wavefront-optimized LASIK for Nearsightedness
Status: Completed | Type: Observational
Sponsor: Edward E. Manche (Other)
Responsible Party: Sponsor-Investigator, Edward E. Manche, Stanford University School of Medicine, Stanford University
Organization: Stanford University (Other)
Other Study IDs: SU-05272010-6188; Stanford Protocol # 18692
Record Dates: First submitted 2010-06-03; First posted 2010-06-07 (Estimated); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Myopia; Astigmatism
Keywords: Wavefront-guided LASIK.; Wavefront-optimized LASIK.; Custom LASIK
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Wavefront-guided LASIK — Wavefront-guided LASIK in one eye using the Allegretto excimer laser
  Other Names: Wavelight Allegretto Eye-Q 400 Hz excimer laser
Procedure: Wavefront-optimized LASIK — Wavefront-optimized LASIK in one eye using the Allegretto excimer laser
  Other Names: Wavelight Allegretto Eye-Q 400 Hz excimer laser

SUMMARY:
The purpose of the study is to compare the results of LASIK surgery when using wavefront-guided excimer laser treatment compared to wavefront optimized excimer laser treatment in patients with nearsightedness with and without astigmatism

DETAILED DESCRIPTION:
This is a research study comparing the outcomes of LASIK surgery for nearsightedness when using the two different excimer laser technologies. Patients will have both eyes treated with the Alcon WaveLight Allegretto excimer laser. You will be one of 150 sighted patients at Stanford to undergo treatment in this clinical research trial. This will be a prospective, randomized, research study in which up to 300 consecutive eyes scheduled to undergo excimer laser in situ keratomileusis (LASIK) using one laser technology in the first eye and the second laser technology in the fellow eye for the correction of myopia (nearsightedness) with or without astigmatism will be enrolled. The choice of which eye receives the wavefront guided technology and which eye receives the wavefront-optimized technology will be randomized prior to enrollment. Randomization will be done according to a randomization schedule. You will know which eye is being treated with which each technology. The randomization will determine only whether your right or left eye is treated with the wavefront guided technology. The other eye will be treated with wavefront-optimized laser technology. You have a fifty percent chance of having your left eye treated with custom wavefront guided technology as your right eye. Subjects will undergo bilateral (both eyes at once) LASIK treatments using the Alcon WaveLight Allegretto excimer laser. All subjects will be followed for one year after the vision correction procedure. Subjects scheduled to undergo LASIK for the correction of myopia (nearsightedness) with or without astigmatism will be screened for eligibility. Eligible subjects will be examined preoperatively to establish a baseline for ocular condition (the general health and glasses prescription of the eyes). Postoperatively, subjects will undergo an ophthalmic evaluation (complete eye examination) at regular intervals as specified in this protocol. Retreatments (a second operation on the same eye for residual nearsightedness) will not be allowed during the first twelve months of this study. If you elect to undergo a retreatment of your LASIK surgery prior to the 12-month post-operative visit, the retreated eye will be exited from the study as of the retreatment date.

Any significant new finding developed during the course of the research which may relate to the subject's willingness to continue participation will be provided to the subject or subject's representative in a timely manner.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 21 and older with healthy eyes.
* Nearsightedness between -7.50 diopters and -7.00 diopters with or without astigmatism of up to 3.50 diopters.

Exclusion Criteria:

* Subjects under the age of 21.
* Patients with excessively thin corneas.
* Patients with topographic evidence of keratoconus.
* Patients with autoimmune diseases.
* Patients who are pregnant or nursing.
* Patients must have similar levels of nearsightedness in each eye. They can not be more than 3.0 diopter of difference between eyes.
* Patients must have similar levels of astigmatism in each eye. They can not have more than 4.0 diopters of difference in nearsightedness or astigmatism between their two eyes.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects age 21 and older with healthy eyes. Nearsightedness between -7.50 diopters and -7.00 diopters with or without astigmatism of up to 3.50 diopters.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2010-04-06 (Actual); Primary Completion 2012-04-30 (Actual); Study Completion 2012-04-30 (Actual)

PRIMARY OUTCOMES:
Changes in best corrected visual acuity | 12 months
Changes in 5 and 25% contrast visual acuity | 12 months
Refractive predictability | 12 months
Uncorrected visual acuity | 12 months

SECONDARY OUTCOMES:
Changes in higher order aberrations | 1 yr
Quality of vision measurement | 1 yr
Topographic analysis | 1 yr

CONTACTS AND LOCATIONS:
Overall Officials: Edward E. Manche, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Result] Sales CS, Manche EE. One-year outcomes from a prospective, randomized, eye-to-eye comparison of wavefront-guided and wavefront-optimized LASIK in myopes. Ophthalmology. 2013 Dec;120(12):2396-2402. doi: 10.1016/j.ophtha.2013.05.010. Epub 2013 Jun 15. PMID 23778091